CLINICAL TRIAL: NCT07302282
Title: The Effectiveness of Pain Neuroscience Education for Patients With Mild to Moderate Carpal Tunnel Syndrome
Brief Title: The Effectiveness of Pain Neuroscience Education for Patients With Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, MAHMUT TALHA SUSAM, MD, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 25-2025/12
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Median Neuropathy; Mononeuropathies; Nerve Compression Syndromes; Education; Exercise; Pain neuroscience education; Carpal tunnel syndrome; Median nerve gliding exercise
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Mononeuropathies; Nerve Compression Syndromes; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: After being diagnosed with mild to moderate CTS based on electrophysiological findings, patients will be randomly assigned to two groups. One group (Group 1) will receive home based exercise program, while the other group (Group 2) will receive home based exercise program and pain neuroscience education.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (home based exercise program) (Active Comparator): Group 1 will receive training on median nerve gliding exercises and self-stretching exercises for the carpal ligament. Patients will be asked to perform 3 sets of median nerve gliding exercises, each consisting of 10 repetitions, and self-stretching exercises for the carpal ligament 3 times a day for 30 seconds as part of home program.
  Interventions: Other: Exercise
- Group 2 (home based exercise program and pain neuroscience education) (Experimental): Group 2 will receive exercise and pain neuroscience education. The exercise will be taught as a home program, similar to the other group. Pain neuroscience training will be provided twice a week for a total of 6 sessions by a trained physical therapist.
  Interventions: Other: Exercise; Behavioral: Pain neuroscience education

INTERVENTIONS:
Other: Exercise — Stretching the transverse carpal ligament helps correct imbalance and provides more space for the median nerve, supporting nerve mobility. Stretching also balances flexor and extensor muscles, reduces tension, and supports overall hand health.
  Nerve gliding exercises, similar to stretching, aim to restore nerve mobility and reduce symptoms.
  Other Names: Median nerve gliding exercises; Self-stretching of carpal ligament
Behavioral: Pain neuroscience education — PNE is an educational intervention aiming to alter a patient's beliefs and cognitions regarding their pain experience. The main contents addressed in the educational session were: neurophysiological aspects of pain, biopsychosocial aspects of pain, concept of peripheral and central sensitization, using audio-visual support, examples and metaphors for a better understanding by the patient, as reported in previous studies.
  Arms: Group 2 (home based exercise program and pain neuroscience education)

SUMMARY:
The goal of this clinical trial is to investigate the effects of Pain Neuroscience Education applied in the treatment of mild and moderate carpal tunnel syndrome (CTS).

The main question it aims to answer is: Does PNE have a therapeutic effect on carpal tunnel syndrome in clinical and ultrasonographic terms? Researchers will compare whether PNE creates a synergistic effect alongside home based exercise programs and splint application in mild to moderate CTS, and will objectively demonstrate potential benefits such as relief from pain and numbness.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is a common compressive neuropathy of the median nerve that presents with symptoms of numbness and tingling in the median nerve distribution of the hand. If symptoms are not treated early, they become chronic. Factors affecting the severity of chronic pain include; biological, psychological and social/environmental etc.

Pain neuroscience education is a treatment strategy that aims to teach patients about the effects of their beliefs and behaviors on the formation of their pain experiences. This education focuses on the role of the central nervous system in pain by raising awareness about the neurobiology and neurophysiology of pain. It focuses on remodelling the behavioral approach to pain perception rather than anatomical damage. This approach aims to reduce patients' fear and catastrophizing by helping them better understand pain. Various metaphors, examples, and visuals are used during PNE to help patients understand pain mechanisms. PNE is thought to have an impact not only on pain but also on disability, functionality, and quality of life. PNE has been documented to have a positive effect not only on pain but also on other important factors such as disability, functionality, and quality of life.

A clinical study has shown that adding PNE to a telerehabilitation program has some positive effects, such as a reduction in symptom severity in patients with carpal tunnel syndrome. However, the number of studies in the literature on the efficacy of PNE in carpal tunnel syndrome is limited to a single study and is based on subjective methods such as patient statements. Unlike the previous study, this study will use objective and innovative assessment methods such as ultrasonography, quantitative sensory test and examination to evaluate symptoms and function.

The evaluation methods used in the study will enable a more in-depth and reliable analysis of symptom management and recovery processes, thereby facilitating the collection of more accurate and reliable data. As there are no similar studies using objective evaluation methods, the methodological contributions of this study will be highly valuable. By offering an innovative approach to pain management and rehabilitation through conservative treatment, it will make significant contributions to both scientific literature and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having a diagnosis of mild or moderate CTS confirmed by ENMG
* Having complaints of pain and numbness in the first three fingers of the hand for at least 3 months

Exclusion Criteria:

* Presence of severe CTS findings on electrophysiological examination
* Presence of metabolic diseases such as uncontrolled diabetes and hypothyroidism
* Presence of inflammatory rheumatic disease (e.g., rheumatoid arthritis)
* Presence of other neuromuscular diseases affecting the hand and wrist (Polyneuropathy, Cervical radiculopathy, peripheral nerve damage, Brachial plexus damage, other entrapment neuropathies, etc.)
* History of hand and wrist trauma
* History of neck and wrist surgery
* History of steroid injection into the carpal tunnel within the last 3 months
* History of physical therapy application to wrist within the last 3 months
* Deformity preventing the use of a splint on the wrist
* Previous participation in a program for the psychological management of chronic pain
* Cognitive dysfunction preventing cooperation with tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire - Symptom Severity Scale | Baseline, in the 3rd week and in the 6th week
  Symptom Severity Scale is an 11-item questionnaire used to assess symptom severity in individuals with CTS. Each item is scored from 1 to 5. Scores range from 1 (no symptoms) to 5 (worst symptoms). The patient's symptom severity score is the average score of 11 items.
Boston Carpal Tunnel Questionnaire - Functional Status Scale | Baseline, in the 3rd week and in the 6th week
  Functional Status Scale is an 8-item questionnaire used to assess the functional status of patients with CTS. Each item is scored from 1 to 5. Scores range from 1 (no functional deficit) to 5 (worst possible function). The patient's functional status score is the average of all 8 items.
Numerical Rating Scale | Baseline, in the 3rd week and in the 6th week
  Patients rate the current pain intensity from 0 ("no pain") to 10 ("worst possible pain").
6-item carpal tunnel syndrome symptom scale (CTS-6) | Baseline, in the 3rd week and in the 6th week
  6 items are evaluated out of a total of 26 points. If the patient's total score is above 5, the probability of carpal tunnel syndrome is 25%, while if it is above 12, the probability reaches 80%.
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | Baseline, in the 3rd week and in the 6th week
  It consists of a total of 7 items. The scale is scored between 0 and 24, with a score of 12 or higher suggesting neuropathic pain.

SECONDARY OUTCOMES:
Ultrasound median nerve cross-sectional area | Baseline, in the 3rd week and in the 6th week
  The cross-sectional area of the median nerve is significantly higher in CTS patients compared to the normal population. Ultrasound, which is used to evaluate the median nerve and determine the underlying etiology, is also used to monitor the effectiveness of the treatment. The cross-sectional area measurement of the median nerve will be recorded in mm².
Semmes-Weinstein Monofilament Test | Baseline, in the 3rd week and in the 6th week
  It is used to assess light touch sensation. The assessment is performed using 5 separate monofilaments. The numerical value in the test kits represents the logarithm of 10 times the force required to bend the monofilament, expressed in milligrams. The numerical values are 2.83 (normal light touch sensation), 3.61 (decreased light touch), 4.31 (decreased protective sensation), 4.56 (loss of protective sensation), and 6.65 (loss of deep pressure sensation). The test is performed by applying the monofilament to the tip of the index finger at a 90-degree angle to the skin for 1.5 seconds, repeated three times. The patient must perceive at least one of the monofilament applications as normal. Failure to perceive the 2.83 threshold value is significant for carpal tunnel syndrome.
Two-Point Discrimination Test (2PD) | Baseline, in the 3rd week and in the 6th week
  It is used to assess cortical tactile sensation. The test is applied to the lateral part of the volar surface of the index finger tip. During the test, patients are asked to close their eyes and indicate whether they feel a single or double point. To prevent incorrect sensory perception, pressure exceeding 1 mm is not applied to the skin. The distance between the two points is increased by 1 mm at a time, starting from 1 mm, until the patient feels two distinct points. In the evaluation, a measurement value perceived as two points is considered normal if it is below 6 mm. The minimum distance between two points that can be distinguished by an individual will be tested three times at 1-minute intervals, and the average value will be recorded in centimeters.
Quantitative sensory evaluation | Baseline, in the 3rd week and in the 6th week
  Starting at 32 °C, the Cold Detection Threshold is cooled at a rate of 1 °C per second, and the patient presses the button when they first feel the cold. For the Heat Detection Threshold, the temperature is heated at a rate of 1 °C per second, and the patient presses the button when they first feel the heat. For the cold pain threshold, it is cooled at a rate of 1 °C per second, and the patient presses the button when they feel cold pain. For the hot pain threshold, it is heated at a rate of 1 °C per second, and the patient presses the button when they feel hot pain. Each measurement is taken 3 times, and the average value is recorded in degrees Celsius.
Hand grip strength measurement | Baseline, in the 3rd week and in the 6th week
  The Baseline® hydraulic hand dynamometer-90 kg (Fabrication Enterprises, White Plains, New York 10602, USA) will be used for hand grip strength measurements. According to the test procedure, three measurements will be taken for hand grip and finger grip strength, with one-minute intervals between each measurement, and the average peak force value will be recorded in kilograms.
Finger pinch strength measurement | Baseline, in the 3rd week and in the 6th week
  The Baseline® hydraulic pinchmeter (Fabrication Enterprises, USA) will be used for pinch force measurements. According to the test procedure, three measurements will be taken for hand grip and finger grip strength, with one-minute intervals between each measurement, and the average peak force value will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Talha Susam, MD, Study Chair — Karamanoglu Mehmetbey University Physical Medicine and Rehabilitation; Mahmut Talha Susam, MD, Principal Investigator — Karamanoglu Mehmetbey University Physical Medicine and Rehabilitation; Aynur Başaran, Prof.MD, Principal Investigator — Karamanoglu Mehmetbey University Physical Medicine and Rehabilitation; Süleyman Gül, PhD, Principal Investigator — Karamanoglu Mehmetbey University Physical Medicine and Rehabilitation; Elif Dilara Durmaz, Pt, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided